CLINICAL TRIAL: NCT04372797
Title: Standardized Instruments to Provide Diagnostic and Prognostic Information in Mild Traumatic Brain Injury (mTBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carey Balaban (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); University of Miami (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Carey Balaban, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY20020032; 0011413765 (Other Grant/Funding Number: Uniformed Services University of the Health Sciences)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Mild Traumatic Brain Injury Participants (Experimental): Males and females from 18-50 years of age who present to a recruitment site within 10 days of injury with a diagnosed concussion that meets all of the following criteria: 1) clear mechanism of injury (i.e., direct or indirect impact to head), 2) Glasgow Coma Scale= 13-15, 3) observed or reported signs (e.g., loss of consciousness, amnesia, or confusion) or symptoms (e.g., headache, dizziness, nausea), and 3) neurosensory symptoms.
  Interventions: Device: Diagnostic test
- Control Participants (Active Comparator): Age- and sex-matched control subjects with minor, non-surgical injuries (e.g., sprains, strains) not requiring hospital admission and no history of mild traumatic brain injury will be recruited from the same study sites.
  Interventions: Device: Diagnostic test

INTERVENTIONS:
Device: Diagnostic test — A battery of oculomotor tests

SUMMARY:
This study will establish the capability of a suite of conventional tests and the Neurolign Dx_100 I-PAS goggle system to reliably and objectively detect mTBI in an acute setting when comparing individuals with mTBI to controls with minor injuries in a similarly stressful environment.

DETAILED DESCRIPTION:
The investigators will employ a comprehensive assessment battery to include vestibular/oculomotor, cognitive, and symptom domains using measures that are consistent with the NIH/NINDS common data elements (CDE) and current military clinical practice guidelines (CPG).

Demographic and health history: Subjects will report medical, concussion and health history at your first visit including medications. Subjects may be asked sensitive personal and family history information. Subjects have the right to not disclose the information requested. This medical and concussion history, as well as your date of clearance/recovery from concussion will be abstracted from the medical record for research purposes.

Neurolign Dx_100 I-PAS testing:

I-PAS testing will be conducted by placing the I-PAS goggles on the head of a patient and asking the patient to follow instructions while a set of tests is performed. Each of these tests simply involves eye motions in response to a target. The I-PAS Goggles are FDA approved for the diagnosis of mTBI. Individuals will undergo a subset of tests from the tests listed below.

Tests: Explanation/eye motion Calibration: Adjusting goggles to focus on eyes Gaze horizontal: Looking right and left Predictive saccade: Looking where a subject knows a light will appear Horizontal random Saccade: Looking right and left Vertical random Saccade: Looking up and down Smooth pursuit horizontal: Following an object right and left smoothly Smooth pursuit vertical: Following an object up and down smoothly Memory Guided saccade: Remembering where an object appeared and looking Self-Paced saccade: Self-generated horizontal saccades Anti-saccade: Looking away from an object that appears (opposite direction horizontally, same magnitude) Optokinetic: Following a moving textured background Visual reaction time: Time required to respond with a button press to a visual target Saccade reaction time: Time required to initiate an eye movement to a visual target Auditory reaction time: Time required to indicate with a button press that an auditory stimulus was heard Subjective visual vertical: Aligning a line to be earth-vertical Subjective visual horizontal: Aligning a line to be earth- horizontal Vergence and pupil tests: Binocular disparity step and sinusoidal pursuit tracking by eye and pupil Light Reflex Tests: Consensual pupillary response to light.

Vestibular/Oculomotor Tests Vestibular/Ocular Motor Screening (VOMS) The VOMS will be used to screen for vestibular and oculomotor symptoms and impairment. The VOMS assesses impairment via patient-reported symptom provocation following each of the following components: 1) smooth pursuit, 2) horizontal and vertical saccades, 3) convergence, 4) horizontal and vertical vestibular ocular reflex (VOR) and 5) visual motion sensitivity (VMS). Patients verbally rate changes in headache, dizziness, nausea and fogginess symptoms compared to their immediate pre-assessment state on a scale of 0 (none) to 10 (severe) following each VOMS assessment, to determine if any domain provokes symptoms. Scores on any VOMS item of 2+ reflects a positive screening cut-off for vestibular or oculomotor impairment (Mucha et al., 2014). Convergence is also assessed in the VOMS using both symptom report and objective measurement of the near point of convergence (NPC averaged across 3 trials. NPC values >5 cm reflect a positive clinical screening cut-off. The VOMS requires limited equipment: a 14 pt font NPC hand held fixation stick, metronome, and a 1 page paper scoring form. The VOMS requires approximately 5 minutes to administer and score.

Dynamic Visual Acuity Test (DVAT) To assess vestibulo-ocular reflex function, the clinical version of the DVAT will be performed. First, the lens-corrected static visual acuity will be assessed using a standard Snellen or LogMAR eye chart. The lowest line that all letters can be read will be recorded. For dynamic visual acuity, the patient will flex their head down 30 deg, then rotate their head in the yaw plane at a frequency of about 2 Hz and amplitude of 20-30 deg. A metronome will be used to set the frequency. Again, the lowest line that all letters can be read will be recorded. A loss of greater than 2 lines suggests an impaired VORThe DVAT takes approximately 5 minutes to administer.

Visual Vertigo Analog Scale (VVAS) The VVAS assesses how much dizziness (0-10 visual analog scale) an individual reports for 9 different activities, such as walking through a supermarket aisle, being in a room with fluorescent lights, going down an escalator, walking over a patterned floor, etc. A positive result occurs when an individual rates at least two of the nine items on the VVAS above zero (VVAS positive). The VVAS takes 5 minutes to administer.

Cognitive Immediate Post-concussion Assessment and Cognitive Testing (ImPACT). ImPACT is a computerized neurocognitive test that includes six modules: 1) verbal memory, 2) design memory, 3) X's and O's, 4) symbol matching, 5) color matching, and 6) three letter memory (ImPACT Applications Inc.). These modules are used to form four composite scores: verbal and visual memory (%), visual motor processing speed (#), and reaction time (RT) (sec). The ImPACT also includes the Post-concussion Symptom Scale (PCSS), which is a 22-item self-reported symptom severity inventory of somatic, cognitive, affective and sleep-related symptoms. The ImPACT test takes 20-30 minutes to administer.

Automated Neuropsychological Assessment Measure (ANAM). The ANAM will be used to assess neurocognitive performance. ANAM is a computerized neurocognitive test that includes eight test modules: 1) code substitution delayed, 2) code substitution, 3) matching to sample, 4) mathematical processing, 5) procedural reaction time, 6) simple reaction time, 7) simple reaction time repeated, and 8) go/no go (ANAM v. 4.3; Vista Life Sciences). These modules are scored based on accuracy, speed, and throughput (accuracy/mean reaction time). The ANAM takes approximately 20 minutes to administer.

Symptoms Modified Balance Error Scoring System (mBESS) The BESS measures postural stability and consists of three stances including feet side by side, a tandem stance, and a single-leg stance on the non-dominant leg. The three stances are performed for 20 sec each, three on a firm surface and three stances on a dynamic (medium density foam) surface. All stances are completed with eyes closed and with hands on the iliac crests. Errors include lifting hands off the iliac crests, opening the eyes, stepping, stumbling, or falling, moving the hip into more than a 30 degree of flexion or abduction, lifting the forefoot or heel, or remaining out of the testing position for more than 5 seconds. Each error equals 1 point, with higher scores indicating worse performance. For the current study, the investigators will use the modified BESS (mBESS) that consists of the three stances performed on the firm surface only. Clinical cut-offs for BESS suggest that a total error score 9 or greater indicates clinical impairment in balance. The mBESS takes approximately 5-6 minutes to administer.

Dizziness Handicap Inventory (DHI) The DHI is a 25-item self-report measure that examines dizziness-related handicap. It has good psychometric properties, is not prone to ceiling or floor effects, has been used in the mTBI population, measures deficits across the spectrum of impairments, activities and participation, and is brief to complete. Each item is categorized into one of three domains: functional, emotional, or physical. It was developed with the help of patients who complained of dizziness and uses a three-item response scale, "yes/sometimes/no" scored as "4/2/0" respectively. The DHI has good internal consistency for the total score ( 0.89). The test-retest reliability is high (r = .97) and it is responsive to change in a vestibular population. The DHI has been validated in individuals with mTBI. The DHI takes approximately 5 minutes to complete.

Neurobehavioral Symptom Inventory (NSI) Per the recommendations of the JPC-8/CRMRP Complex Traumatic Brain Injury Rehabilitation Research Clinical Trial Award, the NSI will be completed by all participants. The NSI is a 22-item (i.e. symptom) scale in which participants rate the severity of symptoms on a 5-point scale (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Very Severe) ranging from 0-60.

Behavioral Symptom Inventory-18 (BSI-18) The BSI-18 is an 18-item symptom inventory that assesses the level of psychological distress during the past 7 days on 18 items. The BSI-18 yields total global severity index ranging from 0-72, as well as somatic, depression, and anxiety sub-scale scores. Any sub-scale T-score >63 is reflective of clinical impairment on that sub-scale. The BSI-18 requires 5 minutes to complete and score.

Pittsburgh Sleep Quality Index (PSQI) The PSQI will be used to assess sleep quality. The PSQI is a self-report measure including 18 items that comprise seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Subscale and global PSQI scores are calculated, with higher scores indicating poorer sleep quality.

Administered Tests

Total test time will be 85-90 minutes per subject and will be conducted in private exam rooms or the concussion research lab:

1. ImPACT/PCSS (20-30 min)
2. VOMS (5 min)
3. DVAT (5 min)
4. VVAS (5 min)
5. mBESS (5 min)
6. DHI (5 min)
7. NSI (5 min)
8. BSI-18 (5 min)
9. PSQI (5 min)
10. ANAM (20 min)
11. Neurolign Dx_100 I-PAS (15-20 min)

mTBI participants will complete 3 visits; Visit 1 within 10 days of injury, Visit 2 11-30 days post-injury, and Visit 3 31 or more days post-injury.

mTBI and control participants will complete their testing at either the UPMC Concussion Clinic in a private exam room or the concussion research lab in a research dedicated environment. No testing will occur in an open, non- confidential, public area.

Control participants will complete 1 visit, completing all of the same assessments with the I-PAS system, surveys, and neurocognitive testing. Testing for Control participants will be completed at the concussion research lab in a confidential, dedicated research setting.

Research Coordinators and Research Assistants and clinical faculty (Co-Is) will complete the above-listed procedures with mTBI and Control participants.

ELIGIBILITY:
Inclusion Criteria:

For the mTBI group, participants must present to a recruitment site within 10 days of injury with a diagnosed concussion that meets all of the following criteria:

1. clear mechanism of injury (i.e., direct or indirect impact to head),
2. Glasgow Coma Scale= 13-15, 3) observed or reported signs (e.g., loss of consciousness, amnesia, or confusion) or symptoms (e.g., headache, dizziness, nausea), and
3. neurosensory symptoms.

For Control group, participants will have minor, non-surgical injuries (e.g., sprains, strains) not requiring hospital admission and no history of mTBI will be recruited from the same study sites.

Exclusion Criteria:

1. History of moderate to severe TBI characterized by any of the following:

   1. Penetrating head trauma
   2. GCS< 13 at the time of injury
   3. Associated with LOC > 30 minutes or amnesia >24 hours
   4. Associated with subdural or epidural hemorrhage
2. mTBI history

   1. mTBI Group - history of mTBI within the last 6 months or experiencing head injury symptoms immediately prior to the current head injury or history of 3 or more mTBIs
   2. Controls - No history of mTBI within the last 12 months and no presence of any mTBI-related symptoms at time of enrollment
3. Presence of severe aphasia
4. History of diagnosed psychiatric disorder (e.g., schizophrenia)
5. Documented neurological disorders (e.g., Epilepsy, stroke, dementia)
6. Pregnancy (females will be asked if they are pregnant)
7. Prior disorders of hearing and balance including:

   1. Meniere's disease
   2. Multiple sclerosis
   3. Vestibular neuritis
   4. Vestibular schwannoma
   5. Sudden sensorineural hearing loss
8. History of tumor of the brain or central nervous system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
I-PAS Predictive Saccade Generation Score | 2 minutes
  First predictive saccade to target in a series. Range:1-24. A lower score is better.
I-PAS Antisaccade Task Error Rate | 2 minutes
  Percent of pro-saccadic errors. Range: 0-100%. A lower score is better.
I-PAS Binocular Disparity Vergence Test | 3 minutes
  Two factor discriminant function classifier for mTBI versus Control subjects
I-PAS Optokinetic Slow Phase Gain Symmetry | 2 min
  Comparison of performance in the right and left direction. Range: 0-100%. Lower value is better
I-PAS Smooth Pursuit Velocity Gain Symmetry | 1 min
  Comparison of performance in the right and left direction. Range: 0-100%. Lower value is better.
Vestibular/Ocular Motor Screening (VOMS) score | 5 minutes
  Patients verbally rate changes in headache, dizziness, nausea and fogginess symptoms compared to their immediate pre-assessment state on a scale of 0 (none) to 10 (severe) following each of the following tasks: 1) smooth pursuit, 2) horizontal and vertical saccades, 3) convergence, 4) horizontal and vertical vestibular ocular reflex (VOR) and 5) visual motion sensitivity (VMS). A near convergence point is also measured. Lower scores are better on each component.
Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) | 25 minutes
  ImPACT is a computerized neurocognitive test that includes six modules: 1) verbal memory, 2) design memory, 3) X's and O's, 4) symbol matching, 5) color matching, and 6) three letter memory (ImPACT Applications Inc.). These modules are used to form four composite scores: verbal and visual memory (%), visual motor processing speed (#), and reaction time (RT) (sec). The ImPACT also includes the Post-concussion Symptom Scale (PCSS), which is a 22-item self-reported symptom severity inventory of somatic, cognitive, affective and sleep-related symptoms. Both composite and item scores are used.
Automated Neuropsychological Assessment Measure (ANAM). | 20 minutes
  ANAM is a computerized neurocognitive test that includes eight test modules: 1) code substitution delayed, 2) code substitution, 3) matching to sample, 4) mathematical processing, 5) procedural reaction time, 6) simple reaction time, 7) simple reaction time repeated, and 8) go/no go (ANAM v. 4.3; Vista Life Sciences). These modules are scored based on accuracy, speed, and throughput (accuracy/mean reaction time). Both composite and item scores are used
Dynamic Visual Acuity Test | 5 minutes
  First, the lens-corrected static visual acuity will be assessed using a standard Snellen or LogMAR eye chart. The lowest line that all letters can be read will be recorded. For dynamic visual acuity, the patient will flex their head down 30 deg, then rotate their head in the yaw plane at a frequency of about 2 Hz and amplitude of 20-30 deg. A metronome will be used to set the frequency. Again, the lowest line that all letters can be read will be recorded. A loss of greater than 2 lines suggests an impaired vestibulo-ocular reflex.
Modified Balance Error Scoring System (mBESS) | 5 minutes
  The BESS measures postural stability and consists of three stances including feet side by side, a tandem stance, and a single-leg stance on the non-dominant leg. The three stances are performed for 20 sec each on a firm surface. All stances are completed with eyes closed and with hands on the iliac crests. Errors include lifting hands off the iliac crests, opening the eyes, stepping, stumbling, or falling, moving the hip into more than a 30 degree of flexion or abduction, lifting the forefoot or heel, or remaining out of the testing position for more than 5 seconds. Each error equals 1 point, with higher scores indicating worse performance.
Neurobehavioral Symptom Inventory (NSI) | 5 minutes
  The NSI is a 22-item (i.e. symptom) scale in which participants rate the severity of symptoms on a 5-point scale (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Very Severe) ranging from 0-60. Both composite and item scores will be analyzed.

SECONDARY OUTCOMES:
Visual Vertigo Analog Scale (VVAS) | 5 minutes
  The VVAS assesses how much dizziness (0-10 visual analog scale) an individual reports for 9 different activities. A rating of at least two of the nine items on the VVAS above zero indicates impairment.
Dizziness Handicap Inventory (DHI) | 5 minutes
  The DHI is a 25-item self-report measure that examines dizziness-related handicap. Both domain summary scores and individual ratings will be used. A low score indicates normal function.
Behavioral Symptom Inventory-18 (BSI-18) | 5 minutes
  The BSI-18 is an 18-item symptom inventory that assesses the level of psychological distress during the past 7 days on 18 items. The BSI-18 yields total global severity index ranging from 0-72, as well as somatic, depression, and anxiety sub-scale scores. Any sub-scale T-score >63 is reflective of clinical impairment on that sub-scale.
Pittsburgh Sleep Quality Index (PSQI) | 5 minutes
  The PSQI will be used to assess sleep quality. The PSQI is a self-report measure including 18 items that comprise seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Subscale and global PSQI scores are calculated, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Carey D Balaban, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - University of Miami, Miami, Florida
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the Uniformed Services University Data Repository, as specified by the award agreement with the University of Pittsburgh.

REFERENCES:
- [Background] Collins MW, Kontos AP, Okonkwo DO, Almquist J, Bailes J, Barisa M, Bazarian J, Bloom OJ, Brody DL, Cantu R, Cardenas J, Clugston J, Cohen R, Echemendia R, Elbin RJ, Ellenbogen R, Fonseca J, Gioia G, Guskiewicz K, Heyer R, Hotz G, Iverson GL, Jordan B, Manley G, Maroon J, McAllister T, McCrea M, Mucha A, Pieroth E, Podell K, Pombo M, Shetty T, Sills A, Solomon G, Thomas DG, Valovich McLeod TC, Yates T, Zafonte R. Statements of Agreement From the Targeted Evaluation and Active Management (TEAM) Approaches to Treating Concussion Meeting Held in Pittsburgh, October 15-16, 2015. Neurosurgery. 2016 Dec;79(6):912-929. doi: 10.1227/NEU.0000000000001447. PMID 27741219
- [Background] Kontos, A.P. and M.W. Collins, Concussion: A clinical profile approach to assessment and treatment. 2018, Washington, DC: American Psychological Association Books
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780
- [Background] Balaban C, Hoffer ME, Szczupak M, Snapp H, Crawford J, Murphy S, Marshall K, Pelusso C, Knowles S, Kiderman A. Oculomotor, Vestibular, and Reaction Time Tests in Mild Traumatic Brain Injury. PLoS One. 2016 Sep 21;11(9):e0162168. doi: 10.1371/journal.pone.0162168. eCollection 2016. PMID 27654131
- [Background] Hoffer ME, Balaban C, Szczupak M, Buskirk J, Snapp H, Crawford J, Wise S, Murphy S, Marshall K, Pelusso C, Knowles S, Kiderman A. The use of oculomotor, vestibular, and reaction time tests to assess mild traumatic brain injury (mTBI) over time. Laryngoscope Investig Otolaryngol. 2017 Apr 12;2(4):157-165. doi: 10.1002/lio2.74. eCollection 2017 Aug. PMID 28894835